CLINICAL TRIAL: NCT05322343
Title: Biobank and Brain Health in Bordeaux. A Population-based Cohort to Study the Biology of Brain and Cognitive Aging in Young Seniors
Brief Title: Biobank and Brain Health in Bordeaux.
Acronym: B-cube
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/34
Record Dates: First submitted 2022-03-10; First posted 2022-04-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Brain; Aging; Cognitive Aging; Immunosenescence; Mental Processes; Mental Disorders; Neurocognitive Disorders; Cognition; Brain Diseases; Dementia; Alzheimer Disease; Mental Health; Behavioral Symptoms; Depression; Anxiety
Keywords: Epidemiologic Methods; Risk factors; Public Health; Environmental Exposure; Exposome; Dietary Exposure; Diet; Food and Nutrition; Nutritional Status; Metabolomics; Systems biology; Environmental Biomarkers; Inflammation Mediators
MeSH Terms: conditions — Mental Disorders; Neurocognitive Disorders; Brain Diseases; Dementia; Alzheimer Disease; Psychological Well-Being; Behavioral Symptoms; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires; Urination; Weights and Measures; Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — blood, urine, saliva, hair, nails and nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective cohort: The general population from the age of 55.
  Interventions: Other: Questionnaires; Other: Fasting blood sampling.; Other: Saliva collection and nasal or nasopharyngeal swab; Other: Urine and stool samples; Other: Hair and a tonenail (or hand nail) sampling; Other: Nasal microbiota; Other: Measurements; Other: Neuroimaging; Other: Medical visit

INTERVENTIONS:
Other: Questionnaires — Participants will complete a series of three questionnaires at the V1 (at home, by a trained interviewer) repeated at V7 for the follow up phase:
  1. A general questionnaire, with collection of general health history and exposure data
  2. A nutritional survey (24-hour recall), that will be repeated by telephone twice at 3-month intervals, at the V4 and V5, V6 visits. and V7, V9, V10 et V11 for the follow-up phase
  3. An evaluation of cognitive performance using a validated computerized battery (Cantab®), completed of neuropsychological tests to evaluate dementia syndromes, depressive symptoms and anxiety.
Other: Fasting blood sampling. — In the morning, during the V2 visit by a nurse at the participant's home. Blood collection will include 8 blood tubes (volume approx.. 35.5 mL), plus 2 additional tubes for 500 participants accepting MRI, for a total volume of blood drawn of 41.5 mL for these participants. For the immunological substudy, a second sample will be taken at a distance (after 4 weeks) for 150 volunteer participants meeting the criteria.
  The blood collection is repeated at V8 during the follow-up phase (21 mL).
Other: Saliva collection and nasal or nasopharyngeal swab — On the day of the V2 visit, the nurse will collect a volume of saliva that has flowed spontaneously for 5 min in a sterile 40-mL polypropylene tube, and a nasal or nasopharyngeal swab using a specific kit.
Other: Urine and stool samples — During the V2 visit, the nurse will collect urine and stool samples collected by the participant in the week preceding the appointment, using the equipment provided and kept in the refrigerator. Stool sampling os repeated at V8 during the follow-up phase.
Other: Hair and a tonenail (or hand nail) sampling — During the V2 visit, the nurse will collect some hair and a toenail sample from the participant, in a dedicated envelope. The hair collection is repeated at V8 during the follow-up phase.
Other: Nasal microbiota — Nasal or nasopharyngeal swab
Other: Measurements — In addition to the samples, anthropometric measurements (weight, height,ead, waist, hip, calf and arm circumferences, subjective evaluation of body shape trajectories over the lifecourse), blood pressure, orthostatic hypotension, walking speed, grip strength, and hearing screening of sarcopenia and Parkinson's syndromes will also be collected by the nurse on the day of the V2 visit. Some of these measures (blood pressure, grip strength, screening of sarcopenia and Parkinson's syndromes) are repeated at V8 during the follow-up visit.
  Analyses may be performed on the biobank samples. These analyses will include metabolite assays (Metabolon®), and may include genotyping for research purposes (without searching for specific genes.
Other: Neuroimaging — A multi-sequence MRI will be performed at the V3 visit. None of the sequences used will require contrast injection. The MRI sequences used will be: a 3D MPRAGE T1-weighted sequence, a T2-weighted sequence (FLAIR), a diffusion EPI sequence, a magnetization transfer sequence, and a resting state functional MRI BOLD sequence. The total duration of the MRI examination will be approximately 50 minutes.
  The MRI will be performed at the Bioimaging Institute on an imager dedicated to research activities (3T Prisma Siemens).During V3 visit, a measurement of skin autofluorescence of advanced glycation products will also be performed
Other: Medical visit — For the participants with cognitive disorders (evaluated by the neuropsychologist during the V1 visit) or Parkinson's syndrome (evaluated by the nurse during the V2 visit),a complementary visit by a neurologist may be proposed in order to specify the etiology of these disorders and to establish a possible diagnosis and etiology.

SUMMARY:
B cube is a new generation cohort to study the determinants and natural history of brain aging, using molecular epidemiology, in a representative sample (N=2000) of the general population from the age of 55 (the approximate age of onset of the first cognitive disorders and a target population particularly receptive to prevention messages). Special interest will be given to nutrition, a promising environmental exposure for prevention.

DETAILED DESCRIPTION:
Cognitive aging and associated pathologies, primarily dementia and its main cause Alzheimer's disease, are a major public health issue. Because of the under-diagnosis of dementia in the population and the very long preclinical phase of these diseases, population-based cohorts are essential to better understand brain aging. With the PAQUID and 3-Cités cohorts, the Bordeaux Population Health Research Center (BPH) has been a world pioneer in population-based studies on aging and dementia, and has thus contributed greatly to a better understanding of age-realted brain diseases. As these cohorts are aging, and in view of the importance of studying the early stages of brain aging, it seems essential to continue our research efforts for the prevention of cognitive aging with the establishment of a new cohort of young seniors. In addition to the population-based design of the study, the representativeness of the cohort appears to be a crucial issue (since population-based cohorts depend on the voluntary participation of healthy individuals, unfavorable exposures and altered health states are often largely under-represented, which reduces the variability of exposures and events, leading to an underestimation of prevalences, a decrease in statistical power and a potential bias in the estimation of associations). Finally, the multifactorial nature of brain ageing pathologies now calls for the replacement of the reductionist approach of risk factors by a more holistic vision of the exposome (defined as all the environmental exposures with which an individual is confronted throughout the lifecourse). The development of an integrated approach of complex, high-dimensional, multi-omics biological data (genomics, transcriptomics, epigenomics, metabolomics, proteomics), applied to various biological matrices, is an indispensable tool to deep phenotyping and to the establishment of a new generation etiological epidemiological research framework in the field of brain aging pathologies.

The Biobank and Brain health in Bordeaux cohort (B cube) will include the completion of a general questionnaire (during the V1 visit), a dietary survey (during the V1, V4 and V5 visits), a computerized cognitive battery (during the V1 visit), a collection of biological material (blood, urine, stool, saliva, hair, nails and nasopharyngeal swab) for the constitution of a biobank (during the V2 biobank visit, 2000 samples of blood, urine, hair, nails and 1000 samples expected for the other fluids/samples) An MRI will be performed in volunteers aged 55 to 70 years (during the V3 visit). Finally, a complementary visit by a medical specialist may be proposed to participants with cognitive disorders or Parkinson's syndrome.

Approximately three years after V1, a follow-up phase is proposed to the participant, comprising a block of 6 visits: a general questionnaire accompanied by a computerized cognitive battery (V7), a dietary survey (V7, V9, V10 and V11), a new collection of biological material (V8) including blood samples and hair (for all participants in the follow-up phase) and stool samples (if sampling had not taken place during V2 and for a subsample of participants at follow-up).

ELIGIBILITY:
Inclusion Criteria:

For the main study:

1. live in Bordeaux metropolitan area,
2. be between 55 and 80 years old (included),
3. selected in terms of socioeconomic level, according to a sampling strategy by age groups and income categories representative of the general population between 55 and 80 years of age
4. be affiliated with the social security system,
5. agree to take a blood sample for the biobank.

For the MRI sub-study: be between 55 and 75 years old (included). Inclusion criteria for the immune response substudy: be 70 years of age or older or participate in the MRI study; agree to take a supplemental blood sample for this substudy.

Exclusion Criteria:

For the main study: persons under guardianship (or more generally under protection), unable to give consent to participate.

For the MRI sub-study: have a contraindication to MRI examination (pacemaker, a valve prosthesis or any other internal electrical/magnetic device; history of neurosurgery or aneurysm; claustrophobia; presence of metal fragments in the eyes, brain or spinal cord).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The general population from the age of 55.
Sampling Method: Probability Sample
Enrollment: 2050 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2030-03-22 (Estimated); Study Completion 2030-03-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants for whom samples are available in the biobank and nutritional and cognitive surveys have been completed. | Inclusion visit
  General questionnaire and a computerized cognitive battery.
Number of participants for whom samples are available in the biobank and nutritional and cognitive surveys have been completed. | week 1
  Collection of biological material for the constitution of a biobank
Number of participants for whom samples are available in the biobank and nutritional and cognitive surveys have been completed. | week 2
  An MRI will be performed in volunteers aged 55 to 70 years.
Number of participants for whom samples are available in the biobank and nutritional and cognitive surveys have been completed. | week 12 and week 24
  Dietary survey

SECONDARY OUTCOMES:
Biobank inventory | Week 1
  of the following biological samples
Cognitive performance, assessed through: non-verbal cognition-Neuropsychological | Inclusion visit and V7 (3 years after inclusion visite)
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Cognitive performance, assessed through: non-verbal cognition - Verbal fluency | Inclusion visit and V7 (3 years after inclusion visite)
  Isaacs' set test (IST)
Cognitive performance, assessed through: non-verbal cognition -Dementia | Inclusion visit and V7 (3 years after inclusion visite)
  Clinical Dementia Rating scale-Sum of Boxes (CDR-SOB)
Cognitive performance, assessed through: non-verbal cognition- Mental | Inclusion visit and V7 (3 years after inclusion visite)
  Mini Mental State Examination (MMSE)
Assement anxiety and depressive symptomatology - Anxiety | Inclusion visit and V7 (3 years after inclusion visite)
  Spielberger State-Trait Anxiety Inventory (STAI)
Assement anxiety and depressive symptomatology - Drepression | Inclusion visit and V7 (3 years after inclusion visite)
  Center for Epidemiological Studies-Drepression scale (CES-D).
Nutrition and Lifestyle evaluated | week 12 and week 24
  at the V4 (4 months after inclusion),V5 (8 mounths after inclusion) and V6 (12 months after inclusion) visits; and V7 (3 years after inclusion), V9 (4 months after v7), V10(8 months after v7) et V11(12 months after v7) for the follow-up phase
Study to the microbiota intestinal, nasal and salivary | Week 1 and V8 (1 month after v7 (3 years after inclusion))
  Heterogeneity and diversity.
Immunosenescence mechanism study | Week 1
  Identification of mechanisms immunosenescence
Cognitive performance, assessed through: non-verbal cognition- Mental | Inclusion visit and V7 (3 years after inclusion visite)
  episodic memory: Free and Cued Selective Reminding test (FCSRT) (Grober & Buschke test in French)
Cognitive performance, assessed through: non-verbal cognition- Mental | Inclusion visit and V7 (3 years after inclusion visite)
  Executive functions: Trail Making tests A and B (TMTA and B)
Incapacity and dependance | Inclusion visit and V7 (3 years after inclusion visite)
  Estriction to mobility (Rosow and Breslow)
Incapacity and dependance | Inclusion visit and V7 (3 years after inclusion visite)
  Instrumental and basic activities of Daily Living (Lawton, Katz)
Incapacity and dependance | Inclusion visit and V7 (3 years after inclusion visite)
  Degree of dependency according to french health insurance system (AG.G.I.R)
Nutrition and Lifestyle evaluated | at the V4 (4 months after inclusion),V5 (8 mounths after inclusion) and V6 (12 months after inclusion) visits; and V7 (3 years after inclusion), V9 (4 months after v7), V10(8 months after v7) et V11(12 months after v7) for the follow-up phase
  Physical activity (International Physical Activity Questionnaire)
Nutrition and Lifestyle evaluated | at the V4 (4 months after inclusion),V5 (8 mounths after inclusion) and V6 (12 months after inclusion) visits; and V7 (3 years after inclusion), V9 (4 months after v7), V10(8 months after v7) et V11(12 months after v7) for the follow-up phase
  other lifestyle factors (smoking and alcohol intakes)

CONTACTS AND LOCATIONS:
Overall Officials: Cécilia SAMIERI, Dr, Principal Investigator — Bordeaux Population Health Researh Center Inserm
Locations (1):
- University Hospital of Bordeaux, Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No